CLINICAL TRIAL: NCT04886635
Title: A Prospective Cohort Study on Active Surveillance After Neoadjuvant Chemoradiation for Oesophageal Cancer: SANO-2 Study
Brief Title: Surgery As Needed for Oesophageal Cancer - 2
Acronym: SANO-2
Status: Recruiting | Type: Observational
Sponsor: Bas P. L. Wijnhoven (Other)
Responsible Party: Sponsor-Investigator, Bas P. L. Wijnhoven, Principal Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL76567.078.21
Record Dates: First submitted 2021-04-28; First posted 2021-05-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cancer of Esophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Active surveillance — Patients will undergo two clinical response evaluations (CREs) after nCRT. During CRE-1 (5-6 weeks) patients will undergo oesophagogastroduodenoscopy (OGD) with bite-on-bite biopsies. During CRE-2 (10-12 weeks) patients will undergo positron emission tomography with computed tomography (PET-CT), endoscopy with bite-on-bite biopsies and endoscopic ultrasonography (EUS) plus fine-needle aspiration (FNA). If cancer is detected, surgery will be performed. Patients with cCR are eligible for active surveillance where regular CREs are performed to detect regrowth of cancer. Delayed oesophagectomy will be offered to patients with highly suspected or profen locoregional regrowth, without distant metastases. The safety and feasibility of active surveillance depends on several factors monitored in the SANO trial. So far, these stopping rules have not been met. In case one of the stopping rules is reached, further inclusion in the SANO-2 study will be stopped and surgical resection is offered.

SUMMARY:
A prospective cohort study on active surveillance after neoadjuvant chemoradiation for oesophageal cancer: SANO-2 study.

DETAILED DESCRIPTION:
An active surveillance approach after completion of neoadjuvant chemoradiotherapy for locally advanced oesophageal cancer is being investigated in the SANO (Surgery As Needed for Oesophageal cancer) trial, that completed patient inclusion in December 2020. First long term results are expected end 2023. Based on current retrospective studies and short term results of the SANO, to date there is no evidence that active surveillance is unsafe. Within the follow-up of the SANO trial, the safety of active surveillance is continuously monitored. Based on a high participation rate (>90%) in the SANO trial and on the view of the Dutch patient federation for cancer of the digestive tract (SPKS) to offer active surveillance as an alternative treatment option in a controlled setting, there is a demand for a tailored surgery approach after neoadjuvant chemoradiotherapy until results of the SANO trial are available. When patients request active surveillance outside the SANO trial, it is of the utmost importance to set up a prospective cohort study (extension study) in order to monitor safety, implementation and effectiveness of active surveillance outside the SANO trial before the final results of the SANO trail are available.

ELIGIBILITY:
Inclusion Criteria:

* Operable patients who are planned to undergo or who recently underwent neoadjuvant chemoradiotherapy according to CROSS followed by surgical resection for histologically proven oesophageal squamous cell carcinoma or adenocarcinoma of the oesophagus or oesophago-gastric junction
* Age ≥18
* Written, voluntary, informed consent.

Exclusion Criteria:

* Non-FDG-avid tumour at baseline PET-CT scan
* Initial treatment with endoscopic resection
* Patients who underwent of who are planned to undergo definitive chemoradiotherapy
* Language difficulty, dementia or altered mental status prohibiting the understanding and giving of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operable patients who are planned to undergo or who recently underwent neoadjuvant chemoradiotherapy according to CROSS followed by surgical resection for histologically proven oesophageal squamous cell carcinoma or adenocarcinoma of the oesophagus or oesophago-gastric junction.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety of active surveillance (including delayed surgery), measured by the number of patients with adverse events | after the procedure/surgery and at least up to 2 years
  Including:
  * Complications from OGD with bite-on-bite biopsies, EUS-FNA and PET-CT
  * Unresectable or incurable (T4b or R2) regrowth
  * Microscopically non-radical (R1) resection
  * Postoperative mortality (90 day- or in-hospital mortality)
  * Postoperative hospital stay of >60 days
  * Postoperative complications, defined by the Esophagectomy Complications Consensus Group (ECCG)
  * Development of distant metastases

SECONDARY OUTCOMES:
Rate of distant and locoregional relapse | at least up to 2 years
  Defined as the proportion of all patients with cCR who develop distant metastases either locoregional relapse
Progression-free survival (PFS) | From cCR until the date of first documented disease progression or date of death from any cause, whichever came first, assessed at least up to 2 years
  Defined as the interval between cCR and the earliest occurrence of disease progression resulting in primarily (or peroperatively) unresectable disease, locoregional regrowth (after completion of therapy), distant dissemination (during or after completion of treatment) or all-cause death
Overall survival (OS) | From cCR until the date of death from any cause, assessed at least up to 2 years
  Patients with cCR at CRE-2, defined from date of diagnosis to date of all-cause death or to last day of follow-up
The proportion of patients in the active surveillance strategy that opted for decision counseling | at least up to 2 years
  Decision counseling is a conversation with a trained physician who can elicit, examine, and discuss the patient's preferences in such a way that the patients are enabled to reflect on all aspects of his/her preference
The proportion of patients that opted for decision counselling as well as the proportion of patients who switched from preferring active surveillance to preferring immediate surgery or vice versa. | at least up to 2 years
Fear of recurrence of cancer | at least up to 2 years
  Assessed with the validated Cancer Worry Scale, including 8 items rated on a 4-point Likert scale ranging from "never" to "almost always." Scores range from 8 to 32. Higher scores indicate more frequent worries about cancer.
Regret of the decision to undergo active surveillance | at least up to 2 years
  Measured by the validated Decision Regret Scale, including 5 items rated on a 5-point Likert scale ranging from 1 ("strongly agree") to 5 ("strongly disagree"). Two of the statements (items 2 and 4) were phrased in the negative direction to avoid yea-saying bias. Scoring consisted of reversing the scores of the 2 negatively phrased items, then taking the mean of the 5 items. These means were converted to a score ranging from 0 to 100 by subtracting 1 and multiplying by 25. A score of 0 means no regret; a score of 100 means high regret.
Regret of the decision to undergo surgery | at least up to 2 years
  Measured by the validated Decision Regret Scale, including 5 items rated on a 5-point Likert scale ranging from 1 ("strongly agree") to 5 ("strongly disagree"). Two of the statements (items 2 and 4) were phrased in the negative direction to avoid yea-saying bias. Scoring consisted of reversing the scores of the 2 negatively phrased items, then taking the mean of the 5 items. These means were converted to a score ranging from 0 to 100 by subtracting 1 and multiplying by 25. A score of 0 means no regret; a score of 100 means high regret.
The proportion of participating patients in the SANO-2 study who meet all eligibility criteria | after the procedure and at least up to 2 years
The proportion of performed diagnostic modalities performed at appropriate time | after the procedure and at least up to 2 years
  According to the SANO-2 study algorithm
The proportion of all performed CREs performed in correct order | after the procedure and at least up to 2 years
  Defined as PET-CT within 1 week followed by combined OGD and EUS
The proportion of all performed endoscopies with at least 4 bite-on-bite biopsies taken | after the procedure and at least up to 2 years
  When taking bite-on-bite biopsies, a second biopsy is taken exactly at the same location of the first biopsy.
The proportion of performed FNA in case of suspected lymph nodes | after the procedure and at least up to 2 years
  Suspected lymph nodes are defined as round, hypoechoic and larger than 5 mm.
The proportion of performed endoscopic reports which are complete | after the procedure and at least up to 2 years
  OGD for anatomical landmarks which should be described, such as locations of the upper and lower tumour boundary, upper oesophageal sphincter, Z-line (where the squamous epithelium of the oesophagus meets the columnar epithelium), oesophagogastric junction (upper border of gastric folds) and diaphragmatic impression.
The number of biopsies taken and quality of the biopsies | after the procedure and at least up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bas Wijnhoven, Dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] Noordman BJ, Spaander MCW, Valkema R, Wijnhoven BPL, van Berge Henegouwen MI, Shapiro J, Biermann K, van der Gaast A, van Hillegersberg R, Hulshof MCCM, Krishnadath KK, Lagarde SM, Nieuwenhuijzen GAP, Oostenbrug LE, Siersema PD, Schoon EJ, Sosef MN, Steyerberg EW, van Lanschot JJB; SANO study group. Detection of residual disease after neoadjuvant chemoradiotherapy for oesophageal cancer (preSANO): a prospective multicentre, diagnostic cohort study. Lancet Oncol. 2018 Jul;19(7):965-974. doi: 10.1016/S1470-2045(18)30201-8. Epub 2018 Jun 1. PMID 29861116
- [Background] Noordman BJ, Wijnhoven BPL, Lagarde SM, Boonstra JJ, Coene PPLO, Dekker JWT, Doukas M, van der Gaast A, Heisterkamp J, Kouwenhoven EA, Nieuwenhuijzen GAP, Pierie JEN, Rosman C, van Sandick JW, van der Sangen MJC, Sosef MN, Spaander MCW, Valkema R, van der Zaag ES, Steyerberg EW, van Lanschot JJB; SANO-study group. Neoadjuvant chemoradiotherapy plus surgery versus active surveillance for oesophageal cancer: a stepped-wedge cluster randomised trial. BMC Cancer. 2018 Feb 6;18(1):142. doi: 10.1186/s12885-018-4034-1. PMID 29409469
- [Derived] van der Zijden CJ, Lagarde SM, Hermus M, Kranenburg LW, van Lanschot JJB, Mostert B, Nuyttens JJME, Oudijk L, van der Sluis PC, Spaander MCW, Valkema MJ, Valkema R, Wijnhoven BPL; SANO-2 study group. A prospective cohort study on active surveillance after neoadjuvant chemoradiotherapy for esophageal cancer: protocol of Surgery As Needed for Oesophageal cancer-2. BMC Cancer. 2023 Apr 10;23(1):327. doi: 10.1186/s12885-023-10747-z. PMID 37038138